CLINICAL TRIAL: NCT05102136
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single-Center Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Ascending Doses of REGN9933, a Monoclonal Antibody Against Factor XI, in Healthy Adult Subjects
Brief Title: Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of REGN9933 in Adult Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R9933-HV-2107; 2021-002568-34 (EudraCT Number)
Record Dates: First submitted 2021-10-19; First posted 2021-11-01 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Healthy Volunteers
Keywords: HV

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous Cohorts (Experimental): Randomized 6:2 to REGN9933 or placebo
  Interventions: Drug: REGN9933; Drug: Placebo
- Subcutaneous Cohorts (Experimental): Randomized 6:2 to REGN9933 or placebo
  Interventions: Drug: REGN9933; Drug: Placebo

INTERVENTIONS:
Drug: REGN9933 — Administered intravenously (IV) or subcutaneous (SC) per the protocol
Drug: Placebo — Placebo to match REGN9933 in same form; placebo administered IV or SC per the protocol

SUMMARY:
The primary objective of the study is to evaluate the safety and tolerability of single doses of REGN9933 in healthy participants

The secondary objectives of the study are to:

* Evaluate the effects of single doses of REGN9933 on intrinsic/common pathway coagulation
* Evaluate the effects of single doses of REGN9933 on extrinsic/common pathway coagulation
* Characterize the drug concentration profiles and pharmacokinetic (PK) following single escalating doses of REGN9933
* Characterize the concentration profiles of total FXI following single escalating doses of REGN9933
* Assess the immunogenicity of single doses of REGN9933

ELIGIBILITY:
Key Inclusion Criteria:

1. Body mass index between 18.0 and 32.5 kilograms/per metered squared (kg/m^2) (inclusive) at the screening visit.
2. Judged by the investigator to be in good health based on medical history, physical examination, vital sign measurements, and electrocardiogram (ECGs) performed at screening and/or prior to administration of initial dose of study drug.
3. Participant is in good health based on laboratory safety testing obtained at the screening visit and/or prior to administration of initial dose of study drug. Note :Participant with suspected or confirmed Gilbert's disease can be enrolled in the study.
4. Normal activated partial thromboplastin time (aPTT), normal prothrombin time (PT), and normal platelet counts at screening period and at day -1 as defined by the local laboratory
5. Hemoglobin value ≥11.0 grams per deciliter (g/dL) for females and ≥12.9 g/dL for males at screening and day -1
6. Negative fecal occult blood test (FOBT) during screening period
7. Normal Bleeding time test (BTT) at day -1 as defined by the study site

Key Exclusion Criteria:

1. History of any major surgical procedure or clinically significant physical trauma, in the opinion of the investigator, that may pose a risk to the subject by study participation.
2. Whole blood donation within the previous 56 days or plasma donation within the previous 7 days prior to screening
3. Pregnant or breastfeeding women
4. History of clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, psychiatric, neurological, or dermatologic disease, as assessed by the investigator
5. Hospitalized for any reason within 30 days of the screening visit.
6. Current smoker or former smoker, including e-cigarettes, who stopped smoking within 12 months prior to the screening visit
7. Confirmed positive drug test result at the screening visit and/or prior to randomization or a history of drug abuse within a year prior to screening.
8. History of alcohol abuse within the last 2 years prior to dosing
9. Positive for human immunodeficiency virus (HIV), hepatitis B, or and/or hepatitis C per protocol resolved hepatitis B infection is not an exclusion.
10. Any malignancy, except for nonmelanoma skin cancer or cervical/anus in situ, that have been resected with no evidence of metastatic disease for 3 years prior to the screening visit
11. Women of child bearing potential (defined as women who are fertile, following menarche until becoming postmenopausal, unless permanently surgically sterile. The only allowed permanent sterilization methods for this study are hysterectomy and/or bilateral oophorectomy.)

Note: Other protocol defined inclusion/exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of treatment emergent adverse events (TEAE) | Until resolution of pharmacodynamic (PD) effects; approximately 36 days

SECONDARY OUTCOMES:
Change from baseline in activated partial thromboplastin time (aPTT) | Until resolution of PD effects; approximately 36 days
Change from baseline in prothrombin time (PT) | Until resolution of PD effects; approximately 36 days
Concentration of REGN9933 in serum | Until resolution of PD effects; approximately 36 days
Change from baseline in total Factor XI (FXI) concentrations | Until resolution of PD effects; approximately 36 days
The incidence of antidrug antibodies (ADAs) to REGN9933 over time | Until resolution of PD effects; approximately 36 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Regeneron Study Site, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, has made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry), has the legal authority to share the data, and has ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at:
  https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/